CLINICAL TRIAL: NCT07249853
Title: Cilostazol for Preventing Delayed Cerebral Ischemia in Aneurysmal Subarachnoid Hemorrhage: A Prospective, Multicenter, Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Cilostazol for Preventing Delayed Cerebral Ischemia in Aneurysmal Subarachnoid Hemorrhage
Acronym: CAPTAIN
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAPTAIN
Record Dates: First submitted 2025-11-14; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: Aneurysmal Subarachnoid Hemorrhage; Cilostazol; Delayed Cerebral Ischemia
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Cilostazol; BID protein, human

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to the following treatment groups at a 1:1 ratio:
  Experimental Group： Within 24 hours after randomization, patients will receive cilostazol 100 mg twice daily for 14 consecutive days, in addition to the standard aSAH treatment.
  Control Group： Within 24 hours after randomization, patients will receive a placebo twice daily (bid) for 14 consecutive days, in addition to the standard aSAH treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cilostazol Group (Experimental): Administer 100 mg cilostazol, twice daily for 14 days and the standard aneurysmal subarachnoid treatment pathway.
  Interventions: Drug: Cilostazol 100 mg BID
- Control Group (Placebo Comparator): Implement placebo 100mg twice daily for 14 days and the standard aneurysmal subarachnoid treatment pathway.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Cilostazol 100 mg BID — Within 24 hours after randomization, patients will receive cilostazol 100 mg twice daily (BID) for 14 consecutive days, in addition to the standard aSAH treatment.
  Arms: Cilostazol Group
Drug: placebo — Within 24 hours after randomization, patients will receive a placebo twice daily (BID) for 14 consecutive days, in addition to the standard aSAH treatment.
  Arms: Control Group

SUMMARY:
The investigators propose to conduct a multicenter randomized trial to test whether cilostazol reduces the incidence of delayed cerebral ischemia (DCI) following aneurysmal subarachnoid hemorrhage (aSAH) and improves patients' neurological prognosis, while assessing its safety.

DETAILED DESCRIPTION:
The investigators propose to conduct a multicenter randomized trial to test the primary hypothesis of whether cilostazol reduces the incidence of delayed cerebral ischemia (DCI) following aneurysmal subarachnoid hemorrhage (aSAH) and improves patients' neurological prognosis, while assessing its safety. The investigators will recruit 316 patients from 30 hospitals in China. Eligibility criteria for the trial participants include Aged 18-80 years. Diagnosed with subarachnoid hemorrhage (SAH) by computed tomography (CT) scan, and the responsible aneurysm is identified by computed tomography angiography (CTA) or digital subtraction angiography (DSA). Received aneurysm coil embolization or craniotomy clipping within 72 hours of symptom onset. Hunt-Hess grade II-IV. No rebleeding or new intracranial hemorrhage is shown on head CT within 6 hours after surgery. Understand and follow the procedures of clinical trial, participate voluntarily and sign the informed consent (the informed consent can be signed voluntarily by the person or guardian). Patients with multiple aneurysms, Modified Rankin Scale (mRS) score ≥ 3 before onset, contraindications to cilostazol use, severe organic diseases and an expected survival time of less than 90 days, severe liver insufficiency or renal insufficiency before randomization, aneurysm treatment requiring the use of other antiplatelet drugs after interventional therapy, receiving treatment with other investigational drugs or device trials currently will be excluded. Patients will be randomly assigned to the experimental group or control group at a 1:1 ratio. Experimental Group patients will receive cilostazol 100 mg twice daily for 14 consecutive days, in addition to the standard aSAH treatment. Control Group patients will receive a placebo twice daily (bid) for 14 consecutive days, in addition to the standard aSAH treatment. The primary study endpoint is incidence of delayed cerebral ischemia (DCI) in patients with aneurysmal subarachnoid hemorrhage (aSAH) within 14±2 days after randomization. Other secondary endpoints include neurological function prognosis at 90±7 days after randomization, incidence of intracranial rebleeding events within 90±7 days after randomization, incidence of other severe bleeding events within 90±7 days after randomization. This trial will provide important information for the development of clinical guidelines for reducing delayed cerebral ischemia (DCI) in patients with aneurysmal subarachnoid hemorrhage (aSAH).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years.
* Diagnosed with subarachnoid hemorrhage (SAH) by computed tomography (CT) scan, and the responsible aneurysm is clearly identified by computed tomography angiography (CTA) or digital subtraction angiography (DSA).
* Received aneurysm coil embolization or craniotomy clipping within 72 hours of symptom onset.
* Hunt-Hess grade II-IV.
* No rebleeding or new intracranial hemorrhage is shown on head CT within 6 hours after surgery.
* Understand and follow the procedures of clinical trial, participate voluntarily and sign the informed consent (the informed consent can be signed voluntarily by the person or guardian)

Exclusion Criteria:

* Multiple aneurysms (>1aneurysms confirmed by CTA/DSA)
* Modified Rankin Scale (mRS) score ≥ 3 before onset
* Patients with contraindications to cilostazol use:

  1. Allergy to cilostazol
  2. Severe heart failure（New York Heart Association (NYHA) Functional Classification Grade III or IV）
  3. Coagulation disorders or systemic bleeding (e.g., hemophilia, gastrointestinal bleeding, hemoptysis, etc.)
  4. Pregnant or lactating women
* Patients with severe organic diseases and an expected survival time of less than 90 days
* Severe liver insufficiency or renal insufficiency before randomization
* Aneurysm treatment requiring the use of other antiplatelet drugs after interventional therapy
* Currently receiving treatment with other investigational drugs or device trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of delayed cerebral ischemia (DCI) | At 14±2 days after randomization
  Delayed cerebral ischemia (DCI) was defined as the occurrence of clinical deterioration, including new-onset focal neurological deficits (e.g., hemiplegia, aphasia, apraxia, hemianopia, or neglect) and/or a decrease in the consciousness (a Glasgow Coma Scale [GCS] score reduction of at least 2 points, either in the total score or any individual subscore), with symptoms lasting for at least 1 hour and not occurring immediately after aneurysm surgery. Other potential causes of clinical deterioration (e.g., hydrocephalus, rebleeding, fever, infection, metabolic disturbance, epilepsy, etc.) were excluded. Alternatively, DCI was defined as the presence of new infarct lesions on follow-up brain CT/MRI that were not detected on the initial admission brain CT or post-operative follow-up brain CT.

SECONDARY OUTCOMES:
Neurological function prognosis | At 90 days after randomization
  The modified Rankin Scale (mRS) score and Glasgow Outcome Scale (GOS) score were evaluated at 90 days after randomization. Favorable outcome was defined as an mRS score of 0-3 (0-3 indicating no disability to moderate disability; 4-6 indicating moderately severe disability to death) and a GOS score of 3-5 (3-5 indicating severe disability to good recovery).
Incidence of intracranial rebleeding events | At 90±7 days after randomization
  Any new intracranial hemorrhage occurring within 90 days after randomization (whether rebleeding in the surgical area or new intracranial hemorrhage events following cilostazol administration), confirmed by comparing non-contrast CT scan results during follow-up with those of the last post-operative non-contrast CT scan before randomization.
Incidence of other severe bleeding events | At 90 days after randomization
  Any new symptomatic intracranial hemorrhage or any new moderate or severe hemorrhage occurring within 90 days after randomization (defined according to the Bleeding Academic Research Consortium [BARC] criteria as hemorrhage requiring endoscopic treatment, surgical intervention, or blood transfusion [Types 2-3] and fatal hemorrhage [Type 5]).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available. Sharing IPD will require IRB approval from Tiantan Hospital and other participating institutes in China.

REFERENCES:
- [Background] SVIN COVID-19 Global SAH Registry. Global impact of the COVID-19 pandemic on subarachnoid haemorrhage hospitalisations, aneurysm treatment and in-hospital mortality: 1-year follow-up. J Neurol Neurosurg Psychiatry. 2022 Jul 28:jnnp-2022-329200. doi: 10.1136/jnnp-2022-329200. Online ahead of print. PMID 35902229
- [Result] Kim BJ, Lee EJ, Kwon SU, Park JH, Kim YJ, Hong KS, Wong LKS, Yu S, Hwang YH, Lee JS, Lee J, Rha JH, Heo SH, Ahn SH, Seo WK, Park JM, Lee JH, Kwon JH, Sohn SI, Jung JM, Navarro JC, Kang DW; PICASSO investigators. Prevention of cardiovascular events in Asian patients with ischaemic stroke at high risk of cerebral haemorrhage (PICASSO): a multicentre, randomised controlled trial. Lancet Neurol. 2018 Jun;17(6):509-518. doi: 10.1016/S1474-4422(18)30128-5. PMID 29778364
- [Result] Suzuki S, Sayama T, Nakamura T, Nishimura H, Ohta M, Inoue T, Mannoji H, Takeshita I. Cilostazol improves outcome after subarachnoid hemorrhage: a preliminary report. Cerebrovasc Dis. 2011;32(1):89-93. doi: 10.1159/000327040. Epub 2011 Jun 11. PMID 21677432
- [Result] Matsuda N, Naraoka M, Ohkuma H, Shimamura N, Ito K, Asano K, Hasegawa S, Takemura A. Effect of Cilostazol on Cerebral Vasospasm and Outcome in Patients with Aneurysmal Subarachnoid Hemorrhage: A Randomized, Double-Blind, Placebo-Controlled Trial. Cerebrovasc Dis. 2016;42(1-2):97-105. doi: 10.1159/000445509. Epub 2016 Apr 13. PMID 27070952
- [Result] Nakatsuka Y, Kawakita F, Yasuda R, Umeda Y, Toma N, Sakaida H, Suzuki H; , on behalf of the Prospective Registry for Searching Mediators of Neurovascular Events After Aneurysmal Subarachnoid Hemorrhage (pSEED) Group. Preventive effects of cilostazol against the development of shunt-dependent hydrocephalus after subarachnoid hemorrhage. J Neurosurg. 2017 Aug;127(2):319-326. doi: 10.3171/2016.5.JNS152907. Epub 2016 Aug 5. PMID 27494819
- [Result] Sugimoto K, Nomura S, Shirao S, Inoue T, Ishihara H, Kawano R, Kawano A, Oka F, Suehiro E, Sadahiro H, Shinoyama M, Oku T, Maruta Y, Hirayama Y, Hiyoshi K, Kiyohira M, Yoneda H, Okazaki K, Dreier JP, Suzuki M. Cilostazol decreases duration of spreading depolarization and spreading ischemia after aneurysmal subarachnoid hemorrhage. Ann Neurol. 2018 Dec;84(6):873-885. doi: 10.1002/ana.25361. Epub 2018 Nov 29. PMID 30341966
- [Result] Qureshi AI, Akhtar IN, Ma X, Lodhi A, Bhatti I, Beall J, Broderick JP, Cassarly CN, Martin RH, Sharma R, Thakkar M, Suarez JI. Effect of Cilostazol in Animal Models of Cerebral Ischemia and Subarachnoid Hemorrhage: A Systematic Review and Meta-Analysis. Neurocrit Care. 2023 Jun;38(3):698-713. doi: 10.1007/s12028-022-01637-6. Epub 2022 Nov 30. PMID 36450971
- [Result] Yamaguchi-Okada M, Nishizawa S, Mizutani A, Namba H. Multifaceted effects of selective inhibitor of phosphodiesterase III, cilostazol, for cerebral vasospasm after subarachnoid hemorrhage in a dog model. Cerebrovasc Dis. 2009;28(2):135-42. doi: 10.1159/000223439. Epub 2009 Jun 5. PMID 19506373
- [Result] Onal MB, Bilginer B, Narin F, Ziyal MI, Soylemezoglu F, Ozgen T. Comparison of intrathecal cilostazol and nimodipine treatments in subarachnoid hemorrhage: an experimental study in rabbits. Acta Neurochir Suppl. 2011;110(Pt 2):43-8. doi: 10.1007/978-3-7091-0356-2_9. PMID 21125444
- [Result] Nishino A, Umegaki M, Fujinaka T, Yoshimine T. Cilostazol attenuates cerebral vasospasm after experimental subarachnoid hemorrhage. Neurol Res. 2010 Oct;32(8):873-8. doi: 10.1179/016164109X12608733393791. Epub 2010 Mar 26. PMID 20350366
- [Result] Boulouis G, Labeyrie MA, Raymond J, Rodriguez-Regent C, Lukaszewicz AC, Bresson D, Ben Hassen W, Trystram D, Meder JF, Oppenheim C, Naggara O. Treatment of cerebral vasospasm following aneurysmal subarachnoid haemorrhage: a systematic review and meta-analysis. Eur Radiol. 2017 Aug;27(8):3333-3342. doi: 10.1007/s00330-016-4702-y. Epub 2016 Dec 21. PMID 28004163
- [Result] Kherallah RY, Khawaja M, Olson M, Angiolillo D, Birnbaum Y. Cilostazol: a Review of Basic Mechanisms and Clinical Uses. Cardiovasc Drugs Ther. 2022 Aug;36(4):777-792. doi: 10.1007/s10557-021-07187-x. Epub 2021 Apr 16. PMID 33860901
- [Result] Werk M, Langner S, Reinkensmeier B, Boettcher HF, Tepe G, Dietz U, Hosten N, Hamm B, Speck U, Ricke J. Inhibition of restenosis in femoropopliteal arteries: paclitaxel-coated versus uncoated balloon: femoral paclitaxel randomized pilot trial. Circulation. 2008 Sep 23;118(13):1358-65. doi: 10.1161/CIRCULATIONAHA.107.735985. Epub 2008 Sep 8. PMID 18779447
- [Result] Kim SG, Hong JM, Kim HY, Lee J, Chung PW, Park KY, Kim GM, Lee KH, Chung CS, Bang OY. Ischemic stroke in cancer patients with and without conventional mechanisms: a multicenter study in Korea. Stroke. 2010 Apr;41(4):798-801. doi: 10.1161/STROKEAHA.109.571356. Epub 2010 Feb 11. PMID 20150545
- [Result] Bedenis R, Stewart M, Cleanthis M, Robless P, Mikhailidis DP, Stansby G. Cilostazol for intermittent claudication. Cochrane Database Syst Rev. 2014 Oct 31;2014(10):CD003748. doi: 10.1002/14651858.CD003748.pub4. PMID 25358850
- [Result] Lee KS, Lee C, Dhillon PS, Kirollos R, Nga VDW, Yeo TT, Henkes H, Arthur AS, Yeo LLL, Bhogal P. Antiplatelet therapy in aneurysmal subarachnoid hemorrhage: an updated meta-analysis. Neurosurg Rev. 2023 Sep 4;46(1):221. doi: 10.1007/s10143-023-02120-2. PMID 37665377
- [Result] Ohkuma H, Suzuki S, Kimura M, Sobata E. Role of platelet function in symptomatic cerebral vasospasm following aneurysmal subarachnoid hemorrhage. Stroke. 1991 Jul;22(7):854-9. doi: 10.1161/01.str.22.7.854. PMID 1830180
- [Result] Rowland MJ, Hadjipavlou G, Kelly M, Westbrook J, Pattinson KT. Delayed cerebral ischaemia after subarachnoid haemorrhage: looking beyond vasospasm. Br J Anaesth. 2012 Sep;109(3):315-29. doi: 10.1093/bja/aes264. PMID 22879655
- [Result] Mayer SA, Aldrich EF, Bruder N, Hmissi A, Macdonald RL, Viarasilpa T, Marr A, Roux S, Higashida RT. Thick and Diffuse Subarachnoid Blood as a Treatment Effect Modifier of Clazosentan After Subarachnoid Hemorrhage. Stroke. 2019 Oct;50(10):2738-2744. doi: 10.1161/STROKEAHA.119.025682. Epub 2019 Aug 9. PMID 31394993
- [Result] Macdonald RL, Higashida RT, Keller E, Mayer SA, Molyneux A, Raabe A, Vajkoczy P, Wanke I, Bach D, Frey A, Marr A, Roux S, Kassell N. Clazosentan, an endothelin receptor antagonist, in patients with aneurysmal subarachnoid haemorrhage undergoing surgical clipping: a randomised, double-blind, placebo-controlled phase 3 trial (CONSCIOUS-2). Lancet Neurol. 2011 Jul;10(7):618-25. doi: 10.1016/S1474-4422(11)70108-9. Epub 2011 Jun 2. PMID 21640651
- [Result] Hoh BL, Ko NU, Amin-Hanjani S, Chou SH-Y, Cruz-Flores S, Dangayach NS, Derdeyn CP, Du R, Hanggi D, Hetts SW, Ifejika NL, Johnson R, Keigher KM, Leslie-Mazwi TM, Lucke-Wold B, Rabinstein AA, Robicsek SA, Stapleton CJ, Suarez JI, Tjoumakaris SI, Welch BG. 2023 Guideline for the Management of Patients With Aneurysmal Subarachnoid Hemorrhage: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2023 Jul;54(7):e314-e370. doi: 10.1161/STR.0000000000000436. Epub 2023 May 22. PMID 37212182
- [Result] Dorhout Mees SM, Rinkel GJ, Feigin VL, Algra A, van den Bergh WM, Vermeulen M, van Gijn J. Calcium antagonists for aneurysmal subarachnoid haemorrhage. Cochrane Database Syst Rev. 2007 Jul 18;2007(3):CD000277. doi: 10.1002/14651858.CD000277.pub3. PMID 17636626
- [Result] Dorhout Mees SM, Kerr RS, Rinkel GJ, Algra A, Molyneux AJ. Occurrence and impact of delayed cerebral ischemia after coiling and after clipping in the International Subarachnoid Aneurysm Trial (ISAT). J Neurol. 2012 Apr;259(4):679-83. doi: 10.1007/s00415-011-6243-2. Epub 2011 Sep 24. PMID 21947244
- [Result] Macdonald RL, Schweizer TA. Spontaneous subarachnoid haemorrhage. Lancet. 2017 Feb 11;389(10069):655-666. doi: 10.1016/S0140-6736(16)30668-7. Epub 2016 Sep 13. PMID 27637674